CLINICAL TRIAL: NCT04636021
Title: Restoring Non-Emergent Cardiovascular Care in the Peri-COVID 19 Era
Brief Title: Restoring Non-Emergent Cardiovascular Care in the Peri- COVID-19 Era
Acronym: RECIPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pinnacle Health Cardiovascular Institute (Network)
Responsible Party: Principal Investigator, William Bachinsky MD, Director, Cardiovascular Research, Pinnacle Health Cardiovascular Institute
Other Study IDs: UPMCP # 20-007
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Corona Virus Infection
Keywords: COVID-19 testing; outpatient procedures
MeSH Terms: conditions — Coronavirus Infections | interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: COVID-19 testing — Pre and post procedure COVID-19 testing for patients undergoing outpatient cardiac procedures.

SUMMARY:
Pre-procedure and Short-Term COVID-19 Testing of Outpatients Undergoing Non-emergent Invasive Cardiovascular Procedures

ELIGIBILITY:
Inclusion Criteria:

• Outpatients undergoing non-emergent invasive cardiac diagnostic, cardiac interventional, peripheral diagnostic, peripheral interventional, structural heart interventional, electrophysiology diagnostic, ablation, or device implantation procedures

Exclusion Criteria:

* Previous positive COVID-19 test result
* Patients with symptoms concerning for COVID-19, including (but not limited to):

Fever > 38˚C, shortness of breath and/or cough in greater severity from baseline, sore throat, anosmia / dysgeusia, vomiting/diarrhea within 24 hours prior to procedure

* Emergent status including (but not limited to) acute coronary syndromes, acute limb ischemia, stroke, need of temporary pacemaker
* Non-outpatient status including (but not limited to) patients evaluated in the hospital, observational unit, or emergency department

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective cardiac procedures in the time of COVID- 19
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who contract COVID-19 while hospitalized for elective outpatient procedures | Through 30 day follow up period

SECONDARY OUTCOMES:
Patient perception of the effect of pre and post procedure COVID-19 testing on risk of contracting COVID-19 while hospitalized for an elective outpatient procedure. | Through 30 day follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No